CLINICAL TRIAL: NCT02070159
Title: Effect of Lower Loading Dose of Prasugrel Compared With Conventional Loading Dose of Clopidogrel and Prasugrel in Korean Coronary Artery Disease Patients Undergoing Coronary Angiography
Brief Title: Prasugrel With Lower Dose - Loading Dose
Acronym: PRELOAD-LD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, MD. Director, Regional Clinical Trial Center. Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRELOAD-LD
Record Dates: First submitted 2014-02-08; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; prasugrel; platelet function tests
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clopidogrel 600 mg (Active Comparator): Patients administer conventional loading dose of clopidogrel 600 mg as active comparators.
  Interventions: Drug: Clopidogrel 600 mg
- Prasugrel 30 mg (Experimental): Patients administer lower loading dose of prasugrel 30 mg.
  Interventions: Drug: Prasugrel 30 mg
- Prasugrel 60 mg (Active Comparator): Patients administer conventional loading dose of prasugrel 60 mg as active comparators.
  Interventions: Drug: Prasugrel 60 mg

INTERVENTIONS:
Drug: Clopidogrel 600 mg — Patients administer 600 mg of clopidogrel as conventional loading dose of clopidogrel
  Other Names: Plavix 600 mg
  Arms: Clopidogrel 600 mg
Drug: Prasugrel 30 mg — Patients administer 30 mg of prasugrel as lower loading dose of prasugrel.
  Other Names: Effient 30 mg
  Arms: Prasugrel 30 mg
Drug: Prasugrel 60 mg — Patients take 60 mg of prasugrel as conventional loading dose of prasugrel.
  Other Names: Effient 60 mg
  Arms: Prasugrel 60 mg

SUMMARY:
Although prasugrel, recently available thienopyridine derivative, exhibits rapid and potent platelet inhibition, concerns of low on-treatment platelet reactivity have been suggested especially in East Asian ethnicities. The investigators compared the effect of lower loading dose of prasugrel with conventional loading dose of clopidogrel and prasugrel.

DETAILED DESCRIPTION:
Although clopidogrel together aspirin has been a backbone of anti-platelet therapy in coronary artery disease patients, clopidogrel has several limitations. It has delayed onset of peak concentration and pharmacodynamic inter-patient response variability resulting in high on-treatment platelet reactivity (HPR). Those demerits are known to be associated with adverse cardiovascular outcomes.

Prasugrel has a more effective metabolism pathway than clopidogrel and exhibits more rapid and potent platelet inhibition. Recent guidelines recommend prasugrel as a first line antiplatelet agent or put precedence over clopidogrel for the patients with acute coronary syndrome. However, there have been concerns of different pharmacodynamic and pharmacokinetic response to prasugrel in East Asian ethnicities.

In addition, lower loading dose of prasugrel exhibited more potent pharmacodynamic effect than clopidogrel 600 mg with comparable efficacy compared to conventional loading dose of prasugrel in healthy Korean subjects.

The investigators compare the antiplatelet effect of lower loading dose of prasugrel 30 mg with conventional loading dose of clopidogrel 600 mg and prasugrel 60 mg in Korean coronary artery disease patients undergoing elective coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years
* Stable or unstable angina
* Planned to undergo elective coronary angiography

Exclusion Criteria:

* Previous history of transient ischemic attack or stroke
* Intracranial neoplasm
* Uncontrolled malignant disease
* History of antiplatelet or anticoagulation treatment within 1 month
* Contraindication to the study drug
* Bleeding diathesis
* Hemoglobin < 10 g/dl
* Platelet count < 100,000/mm3
* Significant renal insufficiency (glomerular filtration rate <60 mL/min/1.73 m2)
* Significant hepatic impairment (Serum liver enzyme or bilirubin > 3 times normal limit)
* Body weight < 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | at 6 hours after administration of study drug. (2 hours for prasugrel groups)
  Platelet reactivity was measured using traditional light transmission aggregometry (LTA), VerifyNow (Accumetrics, San Diego, CA, USA), and multiple electrode aggregometry (MEA, Dynabyte Medical, Munich, Germany).
  The platelet reactivity was measured at 6 hours after study drug administration (after 2 hours for the prasugrel groups).

SECONDARY OUTCOMES:
Percent inhibition | at 6 hours after administration of study drug. (2 hours for prasugrel groups)
  Percent inhibition is calculated using the following fomula: % inhibition = [(baseline reactivity unit - peak reactivity unit) / baseline reactivity unit] × 100.
  Percent inhibition is measured at the time of peak platelet inhibition. The platelet reactivity was measured at 6 hours after study drug administration (after 2 hours for the prasugrel groups).
HPR | at 6 hours after administration of study drug. (2 hours for prasugrel groups)
  The high platelet reactivity (HPR) was defined as the results of LTA ≥ 48% or ≥ 55%, PRU ≥ 242 or ≥ 275, and result of MEA assay ≥ 37 U or 54 U at the time of peak platelet inhibition The platelet reactivity was measured at 6 hours after study drug administration (after 2 hours for the prasugrel groups).
LPR | at 6 hours after administration of study drug. (2 hours for prasugrel groups)
  The low platelet reactivity (LPR) was defined as LTA < 12, PRU < 85, MEA < 19 at the time of peak platelet inhibition.
  The platelet reactivity was measured at 6 hours after study drug administration (after 2 hours for the prasugrel groups).
Bleeding event | 30 days after study drug administration
  Any event related to bleeding including access site bleeding and peri-procedural bleeding based on BARC and ACUITY criteria.
Adverse reaction | 30 days after study drug administration
  Any adverse reaction related to study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- DongA University Hospital, Busan, South Korea

REFERENCES:
- [Background] Kim MH, Zhang HZ, Jung DK. Pharmacodynamic comparisons for single loading doses of prasugrel (30 mg) and clopidogrel (600 mg) in healthy Korean volunteers. Circ J. 2013;77(5):1253-9. doi: 10.1253/circj.cj-12-0783. Epub 2013 Jan 30. PMID 23363643